CLINICAL TRIAL: NCT00676000
Title: Randomized Trial of Interrupted Versus Continuous Vaginal Closure of Anterior Repair With Mesh
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to decrease in Avaulta mesh kit usage & inability to recruit study subjects.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Danielle Patterson, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007p002015
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Pain; Dyspareunia; Surgical Mesh
MeSH Terms: conditions — Pain; Dyspareunia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Interrupted vaginal closure
  Interventions: Procedure: Interrupted vaginal closure
- 2 (Active Comparator): Continuous vaginal closure
  Interventions: Procedure: Continuous vaginal closure

INTERVENTIONS:
Procedure: Interrupted vaginal closure — Horizontal mattress closure of vaginal mucosa over mesh
  Arms: 1
Procedure: Continuous vaginal closure — Running closure of vaginal mucosa over mesh
  Arms: 2

SUMMARY:
Vaginal prolapse is a common condition that is treated with surgical correction. Recently surgeons have been using mesh to augment the repair of vaginal prolapse. Common complications of this surgery include vaginal pain, pain during sex, infection or erosion of the mesh in the vagina. There are different ways to close the vaginal wall over the mesh used in these procedures. Currently, there is no accepted standard method of closing the vaginal wall. The purpose of this study is to find out the best way to close the surgical wound in the vagina. We will compare interrupted closure (separate stitches) to continuous closure (one long, running stitch). We hope to show in our study that one method of closure is better than the other.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for surgery to correct anterior vaginal prolapse with mesh kit

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Mesh exposure | One year

SECONDARY OUTCOMES:
Pain | One year
Dyspareunia | One year

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Patterson, MD, Principal Investigator — Brigham and Women's Hospital